CLINICAL TRIAL: NCT04481438
Title: Effects of Acupunch Exercises on the Frail Older Adults in Long-Term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chia-Pei Chou, Medical doctor, Family Medicine Department, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201900696B0
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Frailty; Exercise
Keywords: Acupunch exercises; Frailty; long-term care facilities
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): exercise group will receive acupunch exercise
  Interventions: Other: Acupunch Exercises
- control group (No Intervention): control group will maintain the regular activities of their original daily lives

INTERVENTIONS:
Other: Acupunch Exercises — The acupunch exercise program was developed based on Jing-Luo theory of tranditional Chinese Medicine. The experiment group will receive Acupunch exercise for 40 minute sessions, 3 times a week, for 24 weeks
  Arms: exercise group

SUMMARY:
Frailty is a complex elderly problem and a precursor of functional degradation in elder adults. The aim of this study will to test the effects of acupunch exercises on the frail older adults in long-term care facilities.

DETAILED DESCRIPTION:
Frailty is a complex elderly problem and a precursor of functional degradation in elder adults. The cause of frailty is multifactorial. Regular exercise intervension could improve frailty condition and general functional fitness. The acupunch exercise program was developed based on Jing-Luo theory of tranditional Chinese Medicine. The aim of this study will to test the effects of acupunch exercises on the frail older adults in long-term care facilities.

ELIGIBILITY:
Inclusion Criteria:

* frail older adults
* aged 65 and above
* had lived in the long-term care facilities more than 3 months

Exclusion Criteria:

* dementia patient
* psychiatric patient
* spinal cord injury patient

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
handgrip strength | 24 weeks
  handgrip strength measured by the Digital Handgrip Dynamometer (in kilograms)
upper limb muscle endurance | 24 weeks
  upper limb muscle endurance measured by the Arm Curl Test in times per 30 seconds
lower limb muscle endurance | 24 weeks
  lower limb muscle endurance measured by the Chair-to-Stand Test in times per 30 seconds
lung function | 24 weeks
  lung function measured by Peak Flow Meter (in liters)
upper body flexibility | 24 weeks
  upper body flexibility measured by the Back Scratch Test( in centimeters)
forward flexion | 24 weeks
  forward flexion measured by the Chair Sit-and-Reach Test( in centimeters)
shoulder joint flexion | 24 weeks
  shoulder joint flexion measured by protractor( in degree)
shoulder joint abduction | 24 weeks
  shoulder joint abduction measured by protractor( in degree)

SECONDARY OUTCOMES:
frailty status | 24 weeks
  evaluated based on the guidelines of the SOF Research Group

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Pei Chou, MD, Study Chair — Chang Gung Memorial Hospital
Locations (10):
- Taiwan (10):
  - Conservation Center, Daliao, Kaohsiung
  - Elderly Care Center, Fongshan District, Kaohsiung
  - Nursing Home, Gangshan, Kaohsiung
  - Nursing Home, Sanmin, Kaohsiung
  - Elderly Care Center, Renwu, Kaohsiung City
  - Citizens' Home, Yanchao, Kaohsiung City
  - Nursing Home, Pingtung City, Pingtung City
  - Nursing Home, Chaozhou, Pingtung
  - Nursing Home, Pingtung City
  - Senior Citizens' Home, Pingtung City

IPD SHARING:
Plan to Share IPD: No
for personal privacy reason

REFERENCES:
- [Result] Hsiao CY, Chen KM, Tsai HY, Huang HT, Cheng YY, Tsai AY. Self-Perceived Health and Sleep Quality of Community Older Adults after Acupunch Exercises. Am J Geriatr Psychiatry. 2018 May;26(5):511-520. doi: 10.1016/j.jagp.2018.01.199. Epub 2018 Jan 31. PMID 29433845
- [Result] Kojima G. Prevalence of Frailty in Nursing Homes: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2015 Nov 1;16(11):940-5. doi: 10.1016/j.jamda.2015.06.025. Epub 2015 Aug 6. PMID 26255709
- [Derived] Chou CP, Chen KM, Tung HT, Belcastro F, Hsu HF. Physical fitness and frailty status of frail older adults in long-term care facilities after acupunch exercises: A cluster-randomized controlled trial. Exp Gerontol. 2022 Jun 15;163:111799. doi: 10.1016/j.exger.2022.111799. Epub 2022 Apr 4. PMID 35390490